CLINICAL TRIAL: NCT05063578
Title: The Minimum Effective Concentration of Lidocaine for Ultrasound-guided Axillary Block for Arterio-venous Fistula Creation Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Hua Chen, Department of Anesthesiology, Far Eastern Memorial Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 110122-F
Record Dates: First submitted 2021-09-08; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant (Experimental)
  Interventions: Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — Different concentration of lidocaine, injected via axillary block for arterio-venous fistula creation surgery

SUMMARY:
The arteriovenous fistula creation (AVF creation) surgery is essential among patients with end stage renal disease who require hemodialysis. The fistula usually locates at forearm, and is created by connecting artery and vein through surgery. Patients undergone hemodialysis through the fistula six weeks later if fistula becoming mature, which means patent vessel diameter and enough flow for hemodialysis. The primary failure rate of arteriovenous fistula creation is about 20% to 40% according to previous research data. Thrombosis is the most common cause of fistula failure, which require surgical intervention after arteriovenous fistula surgery.

Anesthetic technique influences surgical outcome of arteriovenous fistula. General anesthesia, regional anesthesia, and local anesthesia are both wide-used methods. Regional anesthesia with nerve block remains the most popular method for arteriovenous fistula creation. The vessel dilation effect of regional anesthesia helps not only dilatation of artery and vein, but also the fistula itself, and promotes the successful functional dialysis. Various type of nerve block are used as anesthetic method for AVF creation surgery.

People requiring hemodialysis usually have multiple underlying disease involving other major organ such as heart, lung, liver, and the endocrine system. They are more vulnerable to systemic intravenous anesthetic medication. The metabolic rate and pharmacodynamics of local anesthetic may also alter due to multiple systemic disease when compared with healthy adults. The optimal concentration of lidocaine for AVF creation when using axillary block has not yet been studied. This research is conducted for dosing response of different concentration of lidocaine when using axillary block for AVF creation surgery. We aim to investigate the optimal low effective concentration, the MEC90, which defined as 90% of patients can tolerate the operation at this concentration.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I to III
* Operation site : First time undergone surgery

Exclusion Criteria:

* ASA classification IV to V
* Previous operation at surgical site before
* Allergy to local anesthetics
* Infectious state of injection point
* Neuromuscular disease causing preoperative numbness or weakness of extremities
* History of vascular thromboembolism including stroke, pulmonary embolism
* Peripheral neuropathy
* Patient with psychiatric disease
* Coagulopathy, or patient taking anti-coagulant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Minimal effective concentration of lidocaine solution | Before the operation
  To test the sensory and motor blockade after local anesthetics being injected by dermatome testing of upper extremity

SECONDARY OUTCOMES:
Functional Dialysis | six weeks after the operation
  Percentage (%) of patient who under gone hemodialysis via the fistula created

CONTACTS AND LOCATIONS:
Locations (1):
- Chen Yen Hua, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided